CLINICAL TRIAL: NCT06726070
Title: Investigation of Candidate miRNAs as Potential Biomarkers in the Early Diagnosis of Prostate Cancer and Benign Prostate Hyperplasia
Brief Title: Investigation of the Diagnostic Role of miRNAs in PCa and BPH
Status: Completed | Type: Observational
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ali AKKOC, Assoc. Prof. Dr., Alanya Alaaddin Keykubat University
Other Study IDs: 10354421-2020/16-24
Record Dates: First submitted 2024-11-16; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Benign Prostate Hypertrophy(BPH); Prostate Cancer (Adenocarcinoma)
Keywords: prostate cancer; Benign Prostate Hypertrophy(BPH); miRNA; biomarker; PSA
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prostate Cancer: Prostate Cancer Patients
- Benign Prostatic Hyperplasia: Benign prostatic hyperplasia(BPH) patients
- Control: Healthy control

SUMMARY:
Prostate cancer(PCa) is the second most common cause of cancer-related death in men after lung cancer. Diagnostic methods such as measurement of serum Prostate-specific antigen (PSA) levels used in the clinic still cannot distinguish between benign conditions and prostate cancer, and biopsy is essential for the diagnosis of prostate cancer. Due to the high false-positive rate of PSA, many patients are accidentally biopsied, which carries various risks for patients. Therefore, there is a need for new diagnostic methods to support PSA and the identification of reliable biomarkers for early diagnosis.

microRNAs (miRNAs) are short non-coding RNAs that can be detected in body fluids such as urine, blood and serum. In recent years, miRNAs have been nominated as reliable biomarkers that help us make an accurate diagnosis in many diseases, such as cancer. Although various miRNAs have been detected in the sera of prostate cancer patients, there is still little data on which miRNAs can be used as biomarkers.

In this study, investigators aimed to evaluate the expression levels of miR-107, miR-134-5p, miR-149-5p, miR-370-3p and miR-221 in blood as biomarkers capable of distinguishing PCa from benign prostatic hyperplasia (BPH) and will prevent unnecessary biopsies. In addition, they aimed to compare some clinical features such as serum PSA and Gleason Score with serum miRNA levels and determine the relationship between them.

DETAILED DESCRIPTION:
The present study is a prospective study and consists of three work packages. First, clinical evaluations were made and biopsy samples were taken from patients who applied to the urology clinic, had serum PSA levels higher than 4 ng/ML, and were suspected of prostate cancer. Then, a pathological examination of the biopsy samples was performed and the patients were grouped into PCA and BPH. Finally, molecular analyses were performed on blood samples obtained from patients and healthy controls and all obtained data were statistically evaluated.

ELIGIBILITY:
Inclusion Criteria:

* For all groups, between 40-70 years of age.
* Prostate cancer group: Patients with positive digital rectal examination (DRE) results, serum PSA level above 4 ng/mL and a confirmed pathological diagnosis of Prostate cancer.
* BPH group: Patients with a PSA level over 4 ng/mL and a negative DRE result who were clinically and pathologically diagnosed with BPH.
* Control: Healthy volunteers who applied to the urology outpatient clinic for routine check-ups and whose PSA value was below 4 ng/ml.

Exclusion Criteria:

* To have undergone drug therapy or surgery for prostate cancer,
* To have chronic inflammatory or infectious diseases,
* Were hospitalized within the past year for a chronic illness,
* To have another known malignancy,
* Being outside the age limit of 40-70.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Since the study was about prostate cancer, only male patients were included in the study.
Study Population: Patients applying to the Urology Clinic of Alanya Alaaddin Keykubat University Training and Research Hospital.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of miRNA expressions | March 2023
  Five different miRNAs will be evaluated in the study: miR-107, miR-134-5p, miR-149-5p, miR-370-3p and miR-221

CONTACTS AND LOCATIONS:
Overall Officials: Ali AKKOÇ, Study Chair — Alanya Alaaddin Keykubat University
Locations (1):
- Alanya Alaaddin Keykubat University Training and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study included 20 PCa and 17 BPH patients who were clinically and pathologically confirmed, aged between 40 and 70, and had serum PSA levels above 4 ng/mL. Additionally, 20 healthy volunteers were included in the study as the control group.
  The clinical diagnosis of patients included in the study was conducted at the University Training and Research Hospital Urology Outpatient Clinic, with pathological assessments performed in the Pathology Laboratory. miRNA expression analyses were performed using quantitative real-time polymerase chain reaction (qRT- PCR) in peripheral blood samples.
  All statistical analyses were performed using GraphPad Prism-5 (ver.9.0). Analyses were performed using the Kruskal-Wallis rank or Mann Whitney-U test and Spearman's test was used for correlation analysis. The role of miRNAs as biomarkers in PCa was investigated by drawing the receiver operating characteristic (ROC) curves. Statistical significance was taken as p <0.05.
Supporting Information: Study Protocol, SAP
Time Frame: Ethical approval: 13.02.2020; Project start and completion: 01.06.2020-02.03.2023; Patient registration start and completion: 26.01.2021-05.12.2022; The project duration lasted 2 years and 9 months in total.
Access Criteria: IPD and any additional supporting information can be shared with investigators who write about Prostate cancer.

REFERENCES:
- [Background] Puente-Rivera J, De la Rosa Perez DA, Olvera SIN, Figueroa-Angulo EE, Saucedo JGC, Hernandez-Leon O, Alvarez-Sanchez ME. The Circulating miR-107 as a Potential Biomarker Up-Regulated in Castration-Resistant Prostate Cancer. Noncoding RNA. 2024 Aug 24;10(5):47. doi: 10.3390/ncrna10050047. PMID 39311384
- [Background] Shao N, Ma G, Zhang J, Zhu W. miR-221-5p enhances cell proliferation and metastasis through post-transcriptional regulation of SOCS1 in human prostate cancer. BMC Urol. 2018 Mar 5;18(1):14. doi: 10.1186/s12894-018-0325-8. PMID 29506516
- [Background] Su X, Zhang L, Li H, Cheng P, Zhu Y, Liu Z, Zhao Y, Xu H, Li D, Gao H, Zhang T. MicroRNA-134 targets KRAS to suppress breast cancer cell proliferation, migration and invasion. Oncol Lett. 2017 Mar;13(3):1932-1938. doi: 10.3892/ol.2017.5644. Epub 2017 Jan 25. PMID 28454346
- [Background] Pelka K, Klicka K, Grzywa TM, Gondek A, Marczewska JM, Garbicz F, Szczepaniak K, Paskal W, Wlodarski PK. miR-96-5p, miR-134-5p, miR-181b-5p and miR-200b-3p heterogenous expression in sites of prostate cancer versus benign prostate hyperplasia-archival samples study. Histochem Cell Biol. 2021 Mar;155(3):423-433. doi: 10.1007/s00418-020-01941-2. Epub 2020 Dec 17. PMID 33331954
- [Background] Chen Y, Zhao J, Luo Y, Wang Y, Jiang Y. Downregulated expression of miRNA-149 promotes apoptosis in side population cells sorted from the TSU prostate cancer cell line. Oncol Rep. 2016 Nov;36(5):2587-2600. doi: 10.3892/or.2016.5047. Epub 2016 Aug 25. PMID 27573045
- [Background] Nayak B, Khan N, Garg H, Rustagi Y, Singh P, Seth A, Dinda AK, Kaushal S. Role of miRNA-182 and miRNA-187 as potential biomarkers in prostate cancer and its correlation with the staging of prostate cancer. Int Braz J Urol. 2020 Jul-Aug;46(4):614-623. doi: 10.1590/S1677-5538.IBJU.2019.0409. PMID 32213205
- [Background] Foj L, Ferrer F, Serra M, Arevalo A, Gavagnach M, Gimenez N, Filella X. Exosomal and Non-Exosomal Urinary miRNAs in Prostate Cancer Detection and Prognosis. Prostate. 2017 May;77(6):573-583. doi: 10.1002/pros.23295. Epub 2016 Dec 19. PMID 27990656
- [Background] Vanacore D, Boccellino M, Rossetti S, Cavaliere C, D'Aniello C, Di Franco R, Romano FJ, Montanari M, La Mantia E, Piscitelli R, Nocerino F, Cappuccio F, Grimaldi G, Izzo A, Castaldo L, Pepe MF, Malzone MG, Iovane G, Ametrano G, Stiuso P, Quagliuolo L, Barberio D, Perdona S, Muto P, Montella M, Maiolino P, Veneziani BM, Botti G, Caraglia M, Facchini G. Micrornas in prostate cancer: an overview. Oncotarget. 2017 Jul 25;8(30):50240-50251. doi: 10.18632/oncotarget.16933. PMID 28445135

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT06726070/Prot_SAP_ICF_000.pdf